CLINICAL TRIAL: NCT00491270
Title: Bacterial Vaginosis Screening and Treatment to Reduce Infective Complications, Abortion and Preterm Delivery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: Common Sense (Other)
Responsible Party: Commonsense, Commonsense, Cesarea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: F-7-20.6-1 VER-1
Record Dates: First submitted 2007-06-24; First posted 2007-06-26 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Vaginosis, Bacterial; Abortion, Spontaneous; Premature Birth
Keywords: Vaginosis, Bacterial; Abortion, Spontaneous; Premature Birth
MeSH Terms: conditions — Vaginosis, Bacterial; Abortion, Spontaneous; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VS Sense — An applicator to diagnose pH increase above 5.2

SUMMARY:
To determine whether screening of pregnant women with history of previous preterm delivery or with premature contractions for bacterial vaginosis using VS-SENSE, and treatment of positive women will reduce the risk of spontaneous preterm birth.

DETAILED DESCRIPTION:
This is an open-label, comparative, and prospective study. Pregnant women, pregnancy week 26 to 36+6, between the ages 18-45, who were hospitalized in the high risk department, with history of previous preterm delivery and/or with premature contractions. Patient with premature ruptured membrane will be excluded.

In the hospital pregnant women with history of previous preterm delivery or with premature contractions, (participants) will be examined by speculum with no lubricant, The clinician will use the VS-SENSE to sample vaginal secretions and will immediately observe and record the color obtained.Should the VS-SENSE produce positive results the physician will consider giving clindamycin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant subjects, aged 18-45 years, pregnancy week 26 to 36+6, with history of previous preterm delivery or with premature contractions.

Exclusion Criteria:

* Subject with ruptured membranes.
* Subject with signs and symptoms of pelvic inflammatory disease.
* Subject who has used vaginal douching within 12 hours prior to arrival at the hospital.
* Subject who has applied local antiseptic, antibiotic or vaginal treatment within the previous 3 days.
* Subjects who have had sexual intercourse within the last 12 hours.
* Subject with blood in her vaginal secretions.
* Subject is currently participating in another clinical study that may directly or indirectly affect the results of this study.
* Subject is unable or unwilling to cooperate with study procedures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Does screening for BV using VS-SENSE in pregnant women with h/o preterm delivery or with premature contractions, and treatment will reduce or prevent Late miscarriage, preterm birth, preterm PROM, chorioamnionitis, and postpartum endometritis. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, MD, Principal Investigator — Western Galilee Hospital-Nahariya
Locations (1):
- Department of Obstetrics and Gynecology, Nahariya, Israel